CLINICAL TRIAL: NCT07351370
Title: Efficacy of Two Daily - Use CHX Based Mouth Rinses on Microbial Biofilm Accumulation, Gingivitis Development, and Staining: a Randomized Clinical Trial
Brief Title: Efficacy of Two Daily - Use CHX Based Mouth Rinses on Microbial Biofilm Accumulation, Gingivitis Development, and Staining
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dental School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DentalSchool
Record Dates: First submitted 2026-01-04; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Mouthwashes; Chlorhexidine; Dental Plaque; Gingival and Periodontal Disease; Randomized Controlled Trial
MeSH Terms: conditions — Dental Plaque; Periodontal Diseases | interventions — Chlorhexidine; Cetylpyridinium

STUDY DESIGN:
Intervention Model Description: The interventional study model is a single-center, randomized, controlled, double-blind, parallel-design clinical trial spanning over 3 months. It compares the efficacy of two mouth rinses: 1) CHX 0.05% + CPC 0.05% + H2O2 0.8%, and 2) CHX 0.05% + CPC 0.05%, with a placebo. Participants undergo screening, sign consent forms, and receive oral hygiene instructions before being randomly allocated to one of the three groups. They rinse twice daily for 3 months, and oral health parameters are assessed at baseline and monthly intervals. Compliance is monitored, and potential side effects are evaluated. Participants provide feedback via a questionnaire at the trial's end.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blinding study. This means that neither the participants, their caregivers, nor the researchers processing the data or evaluating the results know which participant is receiving which of the three different mouth rinses. Additionally, it seems that the rinses were placed in plastic containers of the same color and labeling, so neither the participants nor the researchers know which container contains which rinse, achieving complete blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- chlorhexidine 0.05% + cetylpyridinium chloride 0.05% and hydrogen peroxide 0.8% (Experimental): Participants rinsed twice daily for 3 months with a mouthwash containing chlorhexidine 0.05% + cetylpyridinium chloride 0.05% and hydrogen peroxide 0.8% , as adjunct to conventional mechanical oral hygiene. All participants received supragingival prophylaxis and oral hygiene reinforcement prior to the intervention.
  Interventions: Drug: chlorhexidine/ cetylpyridinium chloride/ hydrogen peroxide mouthwash
- CHX 0.05% + CPC 0.05% (Experimental): Participants rinsed twice daily for 3 months with a mouthwash containing chlorhexidine 0.05% and cetylpyridinium chloride 0.05% , as adjunct to conventional mechanical oral hygiene. All participants received supragingival prophylaxis and oral hygiene reinforcement prior to the intervention.
  Interventions: Drug: Chlorhexidine/ cetylpyridinium chloride
- placebo mouthwash (Placebo Comparator): Participants rinsed twice daily for 3 months with placebo mouthwash, as adjunct to conventional mechanical oral hygiene. All participants received supragingival prophylaxis and oral hygiene reinforcement prior to the intervention.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: chlorhexidine/ cetylpyridinium chloride/ hydrogen peroxide mouthwash — All participants were instructed to rinse for 3 months for 1 minute twice a day with 15 ml of the provided solution.
  Arms: chlorhexidine 0.05% + cetylpyridinium chloride 0.05% and hydrogen peroxide 0.8%
Drug: Chlorhexidine/ cetylpyridinium chloride — All participants were instructed to rinse for 3 months for 1 minute twice a day with 15 ml of the provided solution
  Arms: CHX 0.05% + CPC 0.05%
Other: Placebo — All participants were instructed to rinse for 3 months for 1 minute twice a day with 15 ml of the provided solution
  Arms: placebo mouthwash

SUMMARY:
Τhe aim of this randomized clinical trial was to investigate the efficacy of two daily mouth rinses containing CHX and different combinations of H2O2 and CPC, when used adjunctive to mechanical oral hygiene, and compare them with a placebo mouth rinse. The primary outcomes evaluated were changes in i) bacterial biofilm accumulation, ii) gingival inflammation, and iii) tooth staining. Secondarily, patient's satisfaction and perspective after the use of these formulations was assessed.

DETAILED DESCRIPTION:
Trial design: This is a single-center, randomized, controlled, double-blind, parallel-design, 3- month clinical trial that compares the effectiveness of two different mouth rinses: 1) CHX 0.05% + CPC 0.05% + H2O2 0.8%, and 2) CHX 0.05% + CPC 0.05% with a placebο mouth rinse containing the same color as CHX mouth rinses but without antimicrobial agents.

Experimental phases: Following patient screening and selection, individuals received written details about the products and the research objectives, and those who volunteered for the study signed a consent form. All participants underwent scaling, air polishing, and received oral hygiene instructions. Patients were instructed to abstained from using any oral rinses for the following two weeks until they entered the trial. The aim of this preparatory phase was to allow only participants with low PI and GI scores (<15%) to take part in the clinical trial. Individuals with PI and GI ≥ 15% were re-enrolled in the two-weeks preparation phase and were reevaluated for suitability to participate in the trial.

After the preparatory phase, baseline (V0) measurements of PI, GI and stain index (SI) were recorded, and subjects were randomly allocated in one of the three following groups based on the different mouth rinse they received to use:

Group 1: CHX 0.05%+ CPC 0.05% + H2O2 0.8%. Group 2: CHX 0.05% + CPC 0.05% Group 3: Placebo

As a double-blind clinical study, neither the periodontist nor the participants are aware of the actual assigned treatment. In case of immediate unblinding of the patient (e.g., serious adverse events), the researcher has obtained opaque identical envelopes containing information regarding the treatment group to which the participant belongs. In the event of unblinding, the date/time and reason for unblinding are recorded in the research database.

All participants were instructed to rinse for 3 months for 1 minute twice a day with 15 ml of the provided solution. They were also instructed to refrain from eating or drinking for at least half an hour after rinsing, and to avoid intake of more than two glasses of coffee, tea or red wine daily.

The oral rinses were placed in opaque plastic containers of the same color, and with a capacity of 1500 ml. The containers were pre-labeled with the individual patient's serial number, so that both the patients and the examiner were unaware of which of the three oral rinses was being used each time.

At the 1-month (V1), 2-months (V2) and 3-months (V3) re-evaluation, PI, GI, and SI, were recorded as described below. In addition, the examiner monitored for potential side effects, and weighed the containers to evaluate patient's compliance. At the end of the trial a questionnaire was given to the participants to assess the patient's perspective on possible secondary effects, such as taste alteration, staining, burning feeling, and irritation.

Clinical measurements

All measurements were performed by the same examiner (periodontist), who was unaware of the group allocation. The following clinical parameters were evaluated:

* PI (Turesky et al. (1970) modification of the Quigley and Hein index (1962))
* Percentages of dental surface covered by dental plaque (PA%) (Pretty et al., 2005, Sagel et al., 2000).
* GI (Löe and Silness (1963))
* SI (Lobene (1968))
* Time of professional mechanical removal at V3

Questionnaire Patients' perception of the product and possible adverse effects were registered in the questionnaire patients had to fill in, in the last visit, by placing a mark in a 10 cm visual analog scale (VAS). (García-Gargallo et al.2017)

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old)
* Presence of at least 24 teeth
* Presence of teeth #23-13 and #43-33
* Gingival Index (GI) ≤30% (Lindhe, 1981)
* No interdental clinical attachment loss (CAL) at ≥2 non-adjacent teeth or buccal/oral CAL ≥3 mm with probing pocket depth (PPD) >3 mm at ≥2 teeth (Tonetti et al., 2019)
* No known allergy to chlorhexidine (CHX), hydrogen peroxide (H₂O₂), or cetylpyridinium chloride (CPC)
* No fixed or removable orthodontic appliances or removable prostheses
* No use of systemic antibiotics within the 3 months prior to the study
* Non-smokers or light smokers (<5 cigarettes/day)
* Non-pregnant and non-lactating women
* Absence of crowns, fixed partial dentures, or class III/IV/V composite restorations covering more than one-third of the crown, and no deep dental caries extending into dentine

Exclusion Criteria:

* Presented with signs of hypersensitivity, severe irritation, or discomfort during the experimental period
* Were not compliant with the experimental protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
change in plaque index (PI) | baseline, 1 month, 2 months and 3 months
  change in dental plaque accumulation assessed using the plaque index (PI)

CONTACTS AND LOCATIONS:
Locations (1):
- NKUA School of Dentistry, Athens, Attica, Greece